CLINICAL TRIAL: NCT05207696
Title: Comparison of the Efficacy of Platelet-rich Fibrin and Connective Tissue Graft in Interdental Papilla Reconstruction: A Retrospective Trial
Brief Title: Comparison of the Efficacy of Platelet-rich Fibrin and Connective Tissue Graft in Interdental Papilla Reconstruction
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Selcen Ozcan Bulut, Asst.Prof, Hacettepe University
Other Study IDs: GO 18/780
Record Dates: First submitted 2021-12-01; First posted 2022-01-26 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: To Evaluate the Efficacy of Platelet-rich Fibrin in Papilla Reconstruction; To Evaluate the Efficacy of Connective Tissue Graft in Papilla Reconstruction
Keywords: connective tissue graft; papilla reconstruction; platelet rich fibrin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Platelet-rich fibrin (PRF): A total of 28 sites from 12 patients who underwent papilla reconstruction with PRF placed with semilunar incision in the maxillary anterior region were included in PRF group. ( Data of 12 patients were included in the study.)
  Interventions: Other: retrospective data analysis
- Connective tissue graft (CTG): A total of 27 sites from 8 patients who underwent papilla reconstruction with CTG placed with semilunar incision in the maxillary anterior region were included in CTG group. (Data of 8 patients were included in the study.)
  Interventions: Other: retrospective data analysis

INTERVENTIONS:
Other: retrospective data analysis — The data of the patients who underwent papilla reconstruction surgery by one of the authors (S.O.B.) using semilunar incision with either PRF or CTG in the maxillary anterior teeth were included in the study. All selected patients had consent for using their data.The data of the patients included in the study were analyzed.(Baseline (BL) and follow-up (T1( first month) , T3 (third month), T6 (sixth month)) clinical data including periodontal evaluations (gingival index (GI), plaque index (PI), papillary bleeding index, pocket depth (PD), keratinized tissue width (KTW), gingival recession), papilla-associated recordings (alveolar crest-interdental contact point (AC-IC), alveolar crest-papilla tip (AC-PT), papilla tip-interdental contact point (PT-IC), papilla height loss (PHL), interdental tissue stroke (ITS) and papilla presence index (PPI)) and patient satisfaction were analyzed.)

SUMMARY:
Aim: To evaluate the efficacy of platelet-rich fibrin (PRF) or connective tissue graft (CTG) in papilla reconstruction (PR) with semilunar incision (SI) technique.

Materials and Methods: A total of 55 sites (27 CTG and 28 PRF) from 20 patients who underwent PR with either PRF or CTG placed with SI in the maxillary anterior region were included in the study. Baseline (BL) and follow-up (T1( first month), T3 (third month), T6 (sixth month)) clinical data including periodontal evaluations (gingival index (GI), plaque index (PI), papillary bleeding index, pocket depth (PD), keratinized tissue width (KTW), gingival recession), papilla-associated recordings (alveolar crest-interdental contact point (AC-IC), alveolar crest-papilla tip (AC-PT), papilla tip-interdental contact point (PT-IC), papilla height loss (PHL), interdental tissue stroke (ITS) and papilla presence index (PPI)) and patient satisfaction were analyzed.

DETAILED DESCRIPTION:
PT-IC was taken as the primary outcome measure. Normal distribution was assessed by histogram and Shapiro-Wilk test. Continuous variables were represented as mean±SD whereas the categorical variables were reported as numbers and percentages. Chi-square test was used for the comparison of the categorical variables. Since the data was normally distributed, Friedman test was used to analyze the time-dependent changes in both groups and the inter-group comparisons were made with Mann-Whitney test. Generalized Estimating Equation was used for analyzing qualitative and quantitative data, time-dependent changes, and the difference between two methods. Data analysis was performed in IBM SPSS Statistics Version 23, and p<0.05 was considered as a significance threshold.

ELIGIBILITY:
Inclusion Criteria:

* All selected patients had consent for using their data.
* The data of the patients who underwent PR surgery by one of the authors (S.O.B.) using SI with either PRF or CTG in the maxillary anterior teeth having contact points,
* at least 2 mm keratinized tissue width (KTW) with probing depth (PD)≤ 3 mm adjacent to the open embrasure were included.
* It was ensured that all baseline (BL) and follow-up data were available and all patients received a comprehensive phase I periodontal treatment prior to the PR procedure.

Exclusion Criteria:

* the patients with systemic problems,
* having medications known to influence the periodontium
* Using tobacco/alcohol
* The relevant regions did not have endodontic problems/needs, caries and history of periodontal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In Hacettepe University Periodontology Department (Jun 2016-Feb 2018), 186 patients treated with PR were scanned and the data of 55 sites (27 CTG and 28 PRF) from 20 patients meeting the criteria were included.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Alveolar crest-Interdental contact point (AC-IC mm) | baseline
  Crestal bone height was measured after administering local anesthesia for each mesiofacial or distofacial test site. UNC-15(HuFriedy, Chicago, IL, USA) periodontal probe was positioned inter-proximally in the gingival sulcus in a corono - apical direction which was parallel to the long axis of the tooth. The probe was advanced apically until it contacted the crest of the alveolar bone. The distance between the crestal bone and interdental contact point was reported as AC-IC . (measurements are in millimeters)
Alveolar crest-Interdental contact point (AC-IC mm) | T1:1st month
  Crestal bone height was measured after administering local anesthesia for each mesiofacial or distofacial test site. UNC-15(HuFriedy, Chicago, IL, USA) periodontal probe was positioned inter-proximally in the gingival sulcus in a corono - apical direction which was parallel to the long axis of the tooth. The probe was advanced apically until it contacted the crest of the alveolar bone. The distance between the crestal bone and interdental contact point was reported as AC-IC . (measurements are in millimeters)
Alveolar crest-Interdental contact point (AC-IC mm) | T3:3rd month
  Crestal bone height was measured after administering local anesthesia for each mesiofacial or distofacial test site. UNC-15(HuFriedy, Chicago, IL, USA) periodontal probe was positioned inter-proximally in the gingival sulcus in a corono - apical direction which was parallel to the long axis of the tooth. The probe was advanced apically until it contacted the crest of the alveolar bone. The distance between the crestal bone and interdental contact point was reported as AC-IC . (measurements are in millimeters)
Alveolar crest-Interdental contact point (AC-IC mm) | T6: 6th month
  Crestal bone height was measured after administering local anesthesia for each mesiofacial or distofacial test site. UNC-15(HuFriedy, Chicago, IL, USA) periodontal probe was positioned inter-proximally in the gingival sulcus in a corono - apical direction which was parallel to the long axis of the tooth. The probe was advanced apically until it contacted the crest of the alveolar bone. The distance between the crestal bone and interdental contact point was reported as AC-IC . (measurements are in millimeters)
Alveolar crest-Papilla tip (AC-PT mm) | baseline
  Crestal bone height was measured after administering local anesthesia for each mesiofacial or distofacial test site. UNC-15(HuFriedy, Chicago, IL, USA) periodontal probe was positioned inter-proximally in the gingival sulcus in a corono - apical direction which was parallel to the long axis of the tooth. The probe was advanced apically until it contacted the crest of the alveolar bone. The distance between the crestal bone and the tip of the interdental papilla was reported as AC-PT. (measurements are in millimeters)
Alveolar crest-Papilla tip (AC-PT mm) | T1:1st month
  Crestal bone height was measured after administering local anesthesia for each mesiofacial or distofacial test site. UNC-15(HuFriedy, Chicago, IL, USA) periodontal probe was positioned inter-proximally in the gingival sulcus in a corono - apical direction which was parallel to the long axis of the tooth. The probe was advanced apically until it contacted the crest of the alveolar bone. The distance between the crestal bone and the tip of the interdental papilla was reported as AC-PT. (measurements are in millimeters)
Alveolar crest-Papilla tip (AC-PT mm) | T3:3rd month
  Crestal bone height was measured after administering local anesthesia for each mesiofacial or distofacial test site. UNC-15(HuFriedy, Chicago, IL, USA) periodontal probe was positioned inter-proximally in the gingival sulcus in a corono - apical direction which was parallel to the long axis of the tooth. The probe was advanced apically until it contacted the crest of the alveolar bone. The distance between the crestal bone and the tip of the interdental papilla was reported as AC-PT. (measurements are in millimeters)
Alveolar crest-Papilla tip (AC-PT mm) | T6: 6th month
  Crestal bone height was measured after administering local anesthesia for each mesiofacial or distofacial test site. UNC-15(HuFriedy, Chicago, IL, USA) periodontal probe was positioned inter-proximally in the gingival sulcus in a corono - apical direction which was parallel to the long axis of the tooth. The probe was advanced apically until it contacted the crest of the alveolar bone. The distance between the crestal bone and the tip of the interdental papilla was reported as AC-PT. (measurements are in millimeters)
Papilla tip-Interdental contact point (PT-IC mm) | baseline
  the periodontal probe was positioned inter-proximally. The distance between interdental contact point and the tip of the interdental papilla was reported as PT-IC. (measurements are in millimeters)
Papilla tip-Interdental contact point (PT-IC mm) | T1:1st month
  the periodontal probe was positioned inter-proximally. The distance between interdental contact point and the tip of the interdental papilla was reported as PT-IC. (measurements are in millimeters)
Papilla tip-Interdental contact point (PT-IC mm) | T3:3rd month
  the periodontal probe was positioned inter-proximally. The distance between interdental contact point and the tip of the interdental papilla was reported as PT-IC. (measurements are in millimeters)
Papilla tip-Interdental contact point (PT-IC mm) | T6: 6th month
  the periodontal probe was positioned inter-proximally. The distance between interdental contact point and the tip of the interdental papilla was reported as PT-IC. (measurements are in millimeters)
Papilla Height Loss (PHL)(Nordland and Tarnow classification system) | baseline
  Each interdental papilla was scored as 0-3 based upon Nordland and Tarnow's classification system The following scores were assigned to the papilla at baseline, T1,T3 and T6. Normal:Interdental papilla fills embrasure space to the apical extent of the interdental contact point/area.
  Class-I. The tip of the interdental papilla lies between the interdental contact point and the most coronal extent of the inter proximal CEJ (the cemento-enamel junction) (space present but inter proximal CEJ is not visible) Class-II.The tip of the interdental papilla lies at or apical to the interproximal CEJ but coronal to the apical extent of the facial CEJ(interproximal CEJ visible) Class-III.The tip of the interdental papilla lies level with or apical to the facial CEJ
Papilla Height Loss (PHL)(Nordland and Tarnow classification system) | T1:1st month
  Each interdental papilla was scored as 0-3 based upon Nordland and Tarnow's classification system The following scores were assigned to the papilla at baseline, T1,T3 and T6. Normal:Interdental papilla fills embrasure space to the apical extent of the interdental contact point/area.
  Class-I. The tip of the interdental papilla lies between the interdental contact point and the most coronal extent of the inter proximal CEJ (the cemento-enamel junction) (space present but inter proximal CEJ is not visible) Class-II.The tip of the interdental papilla lies at or apical to the interproximal CEJ but coronal to the apical extent of the facial CEJ(interproximal CEJ visible) Class-III.The tip of the interdental papilla lies level with or apical to the facial CEJ
Papilla Height Loss (PHL)(Nordland and Tarnow classification system) | T3:3rd month
  Each interdental papilla was scored as 0-3 based upon Nordland and Tarnow's classification system The following scores were assigned to the papilla at baseline, T1,T3 and T6. Normal:Interdental papilla fills embrasure space to the apical extent of the interdental contact point/area.
  Class-I. The tip of the interdental papilla lies between the interdental contact point and the most coronal extent of the inter proximal CEJ (the cemento-enamel junction) (space present but inter proximal CEJ is not visible) Class-II.The tip of the interdental papilla lies at or apical to the interproximal CEJ but coronal to the apical extent of the facial CEJ(interproximal CEJ visible) Class-III.The tip of the interdental papilla lies level with or apical to the facial CEJ
Papilla Height Loss (PHL)(Nordland and Tarnow classification system) | T6: 6th month
  Each interdental papilla was scored as 0-3 based upon Nordland and Tarnow's classification system The following scores were assigned to the papilla at baseline, T1,T3 and T6. Normal:Interdental papilla fills embrasure space to the apical extent of the interdental contact point/area.
  Class-I. The tip of the interdental papilla lies between the interdental contact point and the most coronal extent of the inter proximal CEJ (the cemento-enamel junction) (space present but inter proximal CEJ is not visible) Class-II.The tip of the interdental papilla lies at or apical to the interproximal CEJ but coronal to the apical extent of the facial CEJ(interproximal CEJ visible) Class-III.The tip of the interdental papilla lies level with or apical to the facial CEJ
Interdental Tissue Stroke (ITS) (Jemt's classification system) | baseline
  The following scores were assigned to the papilla at baseline, T1,T3 and T6. Each interdental papilla was scored as 0-3 based upon Jemt's classification system
  Score 0: No papilla is present
  Score 1: Less than half of the height of the papilla is present
  Score 2: Half or more of the height of the papilla is present
  Score 3: The papilla fills up the entire proximal space
Interdental Tissue Stroke (ITS) (Jemt's classification system) | T1:1st month
  The following scores were assigned to the papilla at baseline, T1,T3 and T6. Each interdental papilla was scored as 0-3 based upon Jemt's classification system
  Score 0: No papilla is present
  Score 1: Less than half of the height of the papilla is present
  Score 2: Half or more of the height of the papilla is present
  Score 3: The papilla fills up the entire proximal space
Interdental Tissue Stroke (ITS) (Jemt's classification system) | T3:3rd month
  The following scores were assigned to the papilla at baseline, T1,T3 and T6. Each interdental papilla was scored as 0-3 based upon Jemt's classification system
  Score 0: No papilla is present
  Score 1: Less than half of the height of the papilla is present
  Score 2: Half or more of the height of the papilla is present
  Score 3: The papilla fills up the entire proximal space
Interdental Tissue Stroke (ITS) (Jemt's classification system) | T6: 6th month
  The following scores were assigned to the papilla at baseline, T1,T3 and T6. Each interdental papilla was scored as 0-3 based upon Jemt's classification system
  Score 0: No papilla is present
  Score 1: Less than half of the height of the papilla is present
  Score 2: Half or more of the height of the papilla is present
  Score 3: The papilla fills up the entire proximal space
Papilla presence index (PPI) (by Cardaropoli et al.) | baseline
  The following scores were assigned to the papilla at baseline, T1,T3 and T6. PPI 1: the papilla is completely present and coronally extends to the contact point to completely fill the interproximal embrasure.
  PPI 2: the papilla is no longer completely present and lies apical to the contact point. But the interproximal CEJ (iCEJ) is still not visible.
  PPI 3: the papilla is moved more apical and iCEJ becomes visible. PPI 4: the papilla lies apcal to both iCEJ and buccal CEJ. Each interdental papilla was scored as 1-3 based upon PPI.
Papilla presence index (PPI) (by Cardaropoli et al.) | T1:1st month
  The following scores were assigned to the papilla at baseline, T1,T3 and T6. PPI 1: the papilla is completely present and coronally extends to the contact point to completely fill the interproximal embrasure.
  PPI 2: the papilla is no longer completely present and lies apical to the contact point. But the interproximal CEJ (iCEJ) is still not visible.
  PPI 3: the papilla is moved more apical and iCEJ becomes visible. PPI 4: the papilla lies apcal to both iCEJ and buccal CEJ. Each interdental papilla was scored as 1-3 based upon PPI.
Papilla presence index (PPI) (by Cardaropoli et al.) | T3:3rd month
  The following scores were assigned to the papilla at baseline, T1,T3 and T6. PPI 1: the papilla is completely present and coronally extends to the contact point to completely fill the interproximal embrasure.
  PPI 2: the papilla is no longer completely present and lies apical to the contact point. But the interproximal CEJ (iCEJ) is still not visible.
  PPI 3: the papilla is moved more apical and iCEJ becomes visible. PPI 4: the papilla lies apcal to both iCEJ and buccal CEJ. Each interdental papilla was scored as 1-3 based upon PPI.
Papilla presence index (PPI) (by Cardaropoli et al.) | T6: 6th month
  The following scores were assigned to the papilla at baseline, T1,T3 and T6. PPI 1: the papilla is completely present and coronally extends to the contact point to completely fill the interproximal embrasure.
  PPI 2: the papilla is no longer completely present and lies apical to the contact point. But the interproximal CEJ (iCEJ) is still not visible.
  PPI 3: the papilla is moved more apical and iCEJ becomes visible. PPI 4: the papilla lies apcal to both iCEJ and buccal CEJ. Each interdental papilla was scored as 1-3 based upon PPI.

SECONDARY OUTCOMES:
Gingival index (GI) ( by Löe & Silness 1963) | baseline
  The Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding.
  The GI uses the following scoring system:
  0 = normal gingiva
  1. = mild inflammation: slight change in color, slight edema, no bleeding on probing
  2. = moderate inflammation: redness, edema, and glazing, or bleeding on probing
  3. = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding, ulceration The GI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined.
Gingival index (GI) ( by Löe & Silness 1963) | T1:1st month
  The Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding.
  The GI uses the following scoring system:
  0 = normal gingiva
  1. = mild inflammation: slight change in color, slight edema, no bleeding on probing
  2. = moderate inflammation: redness, edema, and glazing, or bleeding on probing
  3. = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding, ulceration The GI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined.
Gingival index (GI) ( by Löe & Silness 1963) | T3:3rd month
  The Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding.
  The GI uses the following scoring system:
  0 = normal gingiva
  1. = mild inflammation: slight change in color, slight edema, no bleeding on probing
  2. = moderate inflammation: redness, edema, and glazing, or bleeding on probing
  3. = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding, ulceration The GI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined.
Gingival index (GI) ( by Löe & Silness 1963) | T6: 6th month
  The Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding.
  The GI uses the following scoring system:
  0 = normal gingiva
  1. = mild inflammation: slight change in color, slight edema, no bleeding on probing
  2. = moderate inflammation: redness, edema, and glazing, or bleeding on probing
  3. = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding, ulceration The GI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined.
Gingival recession (GR-mm) | baseline
  The distance between buccal CEJ and the most coronal extent marginal gingiva was reported as GR.
  (measurements are in millimeters)
Gingival recession (GR-mm) | T1:1st month
  The distance between buccal CEJ and the most coronal extent marginal gingiva was reported as GR.
  (measurements are in millimeters)
Gingival recession (GR-mm) | T3:3rd month
  The distance between buccal CEJ and the most coronal extent marginal gingiva was reported as GR.
  (measurements are in millimeters)
Gingival recession (GR-mm) | T6: 6th month
  The distance between buccal CEJ and the most coronal extent marginal gingiva was reported as GR.
  (measurements are in millimeters)
Keratinized tissue width (KTW-mm) | baseline
  It extends from the free gingival margin to the mucogingival junction and consists of the free gingiva as well as the attached gingiva. The distance between the most coronal extent free gingiva in buccal and the most coronal extent mucogingival junction was reported as KTW. (measurements are in millimeters)
Keratinized tissue width (KTW-mm) | T1:1st month
  It extends from the free gingival margin to the mucogingival junction and consists of the free gingiva as well as the attached gingiva. The distance between the most coronal extent free gingiva in buccal and the most coronal extent mucogingival junction was reported as KTW. (measurements are in millimeters)
Keratinized tissue width (KTW-mm) | T3:3rd month
  It extends from the free gingival margin to the mucogingival junction and consists of the free gingiva as well as the attached gingiva. The distance between the most coronal extent free gingiva in buccal and the most coronal extent mucogingival junction was reported as KTW. (measurements are in millimeters)
Keratinized tissue width (KTW-mm) | T6: 6th month
  It extends from the free gingival margin to the mucogingival junction and consists of the free gingiva as well as the attached gingiva. The distance between the most coronal extent free gingiva in buccal and the most coronal extent mucogingival junction was reported as KTW. (measurements are in millimeters)
Pocket depth (PD-mm) | baseline
  Periodontal probe was positioned in the gingival sulcus . The distance between the top of the free gingiva and the bottom of the sulcus was reported as PD. (measurements are in millimeters)
Pocket depth (PD-mm) | T1:1st month
  Periodontal probe was positioned in the gingival sulcus . The distance between the top of the free gingiva and the bottom of the sulcus was reported as PD. (measurements are in millimeters)
Pocket depth (PD-mm) | T3:3rd month
  Periodontal probe was positioned in the gingival sulcus . The distance between the top of the free gingiva and the bottom of the sulcus was reported as PD. (measurements are in millimeters)
Pocket depth (PD-mm) | T6: 6th month
  Periodontal probe was positioned in the gingival sulcus . The distance between the top of the free gingiva and the bottom of the sulcus was reported as PD. (measurements are in millimeters)
Plaque index (PI) (by Silness & Löe 1964 ) | baseline
  0- No plaque
  1. -A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. -Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. -Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  The PI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined.
Plaque index (PI) (by Silness & Löe 1964 ) | T1:1st month
  0- No plaque
  1. -A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. -Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. -Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  The PI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined.
Plaque index (PI) (by Silness & Löe 1964 ) | T3:3rd month
  0- No plaque
  1. -A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. -Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. -Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  The PI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined.
Plaque index (PI) (by Silness & Löe 1964 ) | T6: 6th month
  0- No plaque
  1. -A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. -Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. -Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  The PI of the individual can be obtained by adding the values of each tooth and dividing by the number of teeth examined.
Papillary Bleeding Index(PBI) (by Saxer & Muhlemann 1975) | baseline
  The PBI has proven to be particularly useful for assessing inflammation in the interdental papillae by recording bleeding on probing in the interdental areas during the course of treatment.
  Grade 0- no bleeding, normal papilla Grade 1- 20-30 seconds after probing the mesial and distal sulcus with a periodontal probe, a single bleeding point is observed.
  Grade 2- A fine line of blood or several bleeding points become visible at the gingival margin.
  Grade 3- Triangle The interdental triangle becomes more or less filled with blood Grade 4- Immediately after probing, blood flows into the interdental area to cover portions of the tooth and/or gingiva The PBI is calculated by dividing the bleeding number by the total number of papilla examined.
Papillary Bleeding Index(PBI) (by Saxer & Muhlemann 1975) | T1:1st month
  The PBI has proven to be particularly useful for assessing inflammation in the interdental papillae by recording bleeding on probing in the interdental areas during the course of treatment.
  Grade 0- no bleeding, normal papilla Grade 1- 20-30 seconds after probing the mesial and distal sulcus with a periodontal probe, a single bleeding point is observed.
  Grade 2- A fine line of blood or several bleeding points become visible at the gingival margin.
  Grade 3- Triangle The interdental triangle becomes more or less filled with blood Grade 4- Immediately after probing, blood flows into the interdental area to cover portions of the tooth and/or gingiva The PBI is calculated by dividing the bleeding number by the total number of papilla examined.
Papillary Bleeding Index(PBI) (by Saxer & Muhlemann 1975) | T3:3rd month
  The PBI has proven to be particularly useful for assessing inflammation in the interdental papillae by recording bleeding on probing in the interdental areas during the course of treatment.
  Grade 0- no bleeding, normal papilla Grade 1- 20-30 seconds after probing the mesial and distal sulcus with a periodontal probe, a single bleeding point is observed.
  Grade 2- A fine line of blood or several bleeding points become visible at the gingival margin.
  Grade 3- Triangle The interdental triangle becomes more or less filled with blood Grade 4- Immediately after probing, blood flows into the interdental area to cover portions of the tooth and/or gingiva The PBI is calculated by dividing the bleeding number by the total number of papilla examined.
Papillary Bleeding Index(PBI) (by Saxer & Muhlemann 1975) | T6: 6th month
  The PBI has proven to be particularly useful for assessing inflammation in the interdental papillae by recording bleeding on probing in the interdental areas during the course of treatment.
  Grade 0- no bleeding, normal papilla Grade 1- 20-30 seconds after probing the mesial and distal sulcus with a periodontal probe, a single bleeding point is observed.
  Grade 2- A fine line of blood or several bleeding points become visible at the gingival margin.
  Grade 3- Triangle The interdental triangle becomes more or less filled with blood Grade 4- Immediately after probing, blood flows into the interdental area to cover portions of the tooth and/or gingiva The PBI is calculated by dividing the bleeding number by the total number of papilla examined.
Patient-based variables | T1:1st month
  Evaluation was made using the Visual Analog Scale( VAS- 0-10). The experienced pain values, the aesthetic expectations , The gained aesthetics / difficulty variables. these three criteria were evaluated together ( patient satisfaction )
Patient-based variables | T3:3rd month
  Evaluation was made using the Visual Analog Scale( VAS- 0-10). The experienced pain values, the aesthetic expectations , The gained aesthetics / difficulty variables. these three criteria were evaluated together ( patient satisfaction )
Patient-based variables | T6: 6th month
  Evaluation was made using the Visual Analog Scale( VAS- 0-10). The experienced pain values, the aesthetic expectations , The gained aesthetics / difficulty variables. these three criteria were evaluated together ( patient satisfaction )

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Dentistry, Periodontology Department, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma E, Sharma A, Singh K. The role of subepithelial connective tissue graft for reconstruction of interdental papilla: Clinical study. Singapore Dent J. 2017 Dec;38:27-38. doi: 10.1016/j.sdj.2017.05.001. PMID 29229072
- [Background] Singh D, Jhingran R, Bains VK, Madan R, Srivastava R. Efficacy of Platelet-rich Fibrin in Interdental Papilla Reconstruction as Compared to Connective Tissue Using Microsurgical Approach. Contemp Clin Dent. 2019 Oct-Dec;10(4):643-651. doi: 10.4103/ccd.ccd_936_18. PMID 32792824
- [Background] Carnio J, Carnio AT. Papilla reconstruction: Interdisciplinary consideration for clinical success. J Esthet Restor Dent. 2018 Nov;30(6):484-491. doi: 10.1111/jerd.12411. Epub 2018 Sep 8. PMID 30195268